CLINICAL TRIAL: NCT03210818
Title: Effects of Adjustment of Blood Flow of Venoarterial Extracorporeal Membrane Oxygenation Life Support on Microcirculation
Brief Title: Effects of Blood Flow of Venoarterial Extracorporeal Membrane Oxygenation Life Support on Microcirculation
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201703011RINA
Record Dates: First submitted 2017-07-02; First posted 2017-07-07 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2018-07

CONDITIONS: Circulatory Failure
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Extra-corporeal membrane oxygenation life support — Adjustment of blood flow of extra-corporeal membrane oxygenation life support

SUMMARY:
Extra-corporeal membrane oxygenation (ECMO) life support system can provide both cardiac and respiratory support to patients with heart and respiratory failure. It can save time for these patients to regain organ function or to receive transplantation. Both the investigators' team and Ince et al. from the Netherland found that the microcirculatory dysfunction is more severe in ECMO non-survivors. The next step of research is to find out the key factors that affect microcirculation in ECMO patients. Because the blood flow supplied by the venoarterial ECMO (VA-ECMO) is directly related to macrocirculation, this study aims to investigate the effect of adjustment of VA-ECMO blood flow on microcirculation. The investigators hope that the results of this study can help the medical team to improve the quality of ECMO care.

DETAILED DESCRIPTION:
After evaluation, explanation, and acquisition of agreement, the sublingual microcirculation will be examined within 24 h and at 48 h after placement of VA-ECMO. The VA-ECMO blood flow will be recorded, and the baseline microcirculation will be examined. After the ECMO technician adjusting the ECMO flow, sublingual microcirculation will be examined 2 minutes after each adjustment, and the change of ECMO blood flow will be recorded. When the ECMO team plans to weaning off the ECMO within 72 h, the sublingual microcirculation will be examined. The VA-ECMO blood flow will be reduced by ECMO technician, and sublingual microcirculation will be examined 2 minutes after each adjustment of the blood flow. The ECMO parameters, medications, and clinical data will be recorded, and the prognosis will be followed up on the 28th day.

ELIGIBILITY:
Inclusion Criteria:

* Patients who require venoarterial extra-corporeal membrane oxygenation (ECMO) life support

Exclusion Criteria:

* who can not take an examination of sublingual microcirculation within 24 hours after placement of venoarterial ECMO support
* Non-native speakers

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who require venoarterial extra-corporeal membrane oxygenation (ECMO) life support
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-11-05 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Perfused small vessel density | Difference of PSVD between before and after adjustment of VA-ECMO blood flow within 24 hours after placement of VA-ECMO
  Perfused small vessel density [PSVD] measured by incident dark field video microscope

SECONDARY OUTCOMES:
Perfused small vessel density | Difference of PSVD between before and after adjustment of VA-ECMO blood flow on day 2 after placement of VA-ECMO
  Perfused small vessel density [PSVD] measured by incident dark field video microscope
Perfused small vessel density | Difference of PSVD between before and after adjustment of VA-ECMO blood flow within anticipated 72 hours before removal of VA-ECMO
  Perfused small vessel density measured by incident dark field video Perfused small vessel density [PSVD] measured by incident dark field video
Total small vessel density | Difference of TSVD between before and after adjustment of VA-ECMO blood flow within 24 hours after placement of VA-ECMO
  Total small vessel density [TSVD] measured by incident dark field video microscope
Proportion of perfused vessel | Difference of PPV between before and after adjustment of VA-ECMO blood flow within 24 hours after placement of VA-ECMO
  Proportion of perfused vessel (PPV): TSVD/PSVD X 100

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chang Yeh, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No